CLINICAL TRIAL: NCT00000835
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blind Trial to Evaluate the Safety and Immunogenicity of an HIV-1 Pseudovirion Vaccine
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: AVEG 025; 11541 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

SUMMARY:
The purpose of this trial is to determine the safety and immunogenicity of an HIV-1 pseudovirion vaccine given at one antigen dose alone and in combination with each of two different adjuvants using two immunization schedules.

The pseudovirions are virus-like particles generated by in vitro production of HIV-1 viral proteins which are capable of assembly into particles. The presence of gag gene products in addition to envelope glycoprotein should assist in humoral and cellular immunologic responses to internal HIV-1 viral proteins. The pseudovirion vaccine has been tested in preclinical trials in mice, guinea pigs, rabbits, and nonhuman primates with good safety and immunogenicity profile.

DETAILED DESCRIPTION:
The pseudovirions are virus-like particles generated by in vitro production of HIV-1 viral proteins which are capable of assembly into particles. The presence of gag gene products in addition to envelope glycoprotein should assist in humoral and cellular immunologic responses to internal HIV-1 viral proteins. The pseudovirion vaccine has been tested in preclinical trials in mice, guinea pigs, rabbits, and nonhuman primates with good safety and immunogenicity profile.

A total of 78 volunteers will be recruited and randomly assigned to receive pseudovirion vaccine and/or the placebo/adjuvant. All volunteers will receive injections intramuscularly at 0, 1, 3, 6, and 12 months.

Group I (30 volunteers): pseudovirion vaccine w/adjuvant or w/o adjuvant. Group II (30 volunteers): pseudovirion vaccine w/adjuvant or w/o adjuvant. Group III (18 volunteers): adjuvant (QS21 or alum) or saline placebo. NOTE: Group I will receive appropriate adjuvant or saline placebo at Month 3 without pseudovirion vaccine.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Negative ELISA for HIV-1 antibody within 8 weeks of initial immunization.
* CD4 count >= 400 cells/mm3.
* Negative Hepatitis B surface antigen.
* Normal history and physical examination.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and symptoms are excluded:

* Medical or psychiatric condition or occupational responsibilities preclude compliance with the protocol.
* Present psychosis.
* Active syphilis (eligible if serology documented to be a false positive or due to remote, i.e., > 6 months treated infection).
* Active tuberculosis (eligible if positive purified protein derivative test and normal chest x-ray showing no evidence of TB and not requiring isoniazid therapy).
* Hepatitis B antigenemia.

Concurrent Medication:

Excluded:

Immunosuppressive medications.

Patients with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, malignancy, or autoimmune disease.
* History of cancer unless there has been surgical excision followed by sufficient observation period to give a reasonable assurance of cure.
* History of suicide attempts, recent suicidal ideation or who have past psychosis.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care (e.g. Stevens-Johnson syndrome, bronchospasm, or hypotension).

Prior Medication:

Excluded:

* Prior receipt of HIV-1 vaccines or placebo recipient in a previous HIV vaccine trial.
* Use of experimental agents within 30 days prior to study.
* Live attenuated vaccines within 60 days of study.
* Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) within 2 weeks prior to study.

Prior Treatment:

Excluded:

Receipt of blood products or immunoglobulin in the past 6 months.

Risk Behavior:

Excluded:

Volunteers having identifiable higher risk behavior for HIV infection as determined by screening questions designed to identify risk factors for HIV infection, specifically:

* History of injection drug use within the last 12 months prior to enrollment.
* Higher or intermediate risk sexual behavior as defined by the AVEG ( i.e., meeting the criteria for AVEG Risk Group C or D).

Volunteers risk behavior for HIV infection will be determined upon information obtained from a questionnaire and from the AIDS Vaccine Evaluation Group (AVEG) risk behavior guidelines.

NOTE:

* Only those volunteers meeting the criteria for AVEG Risk Groups A and B will be enrolled in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gorse G, Study Chair